CLINICAL TRIAL: NCT01209702
Title: A Ph II/III Seamless, Multi-center, Randomized, Double-blind, Placebo-controlled Study of the Reduction in Signs and Symptoms and Inhibition of Structural Damage During Treatment With Tocilizumab Versus Placebo in Patients With Ankylosing Spondylitis Who Have Failed Non-steroidal Anti-inflammatory Drugs and Are naïve to TNF Antagonist Therapy NSAIDs
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Patients With Ankylosing Spondylitis Who Have Failed Treatment With NSAIDs
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment halted: Failed to achieve efficacy
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA22823; 2009-017443-34
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Part 1: Placebo (Placebo Comparator): Participants received intravenous infusions of placebo once every 4 weeks until Week 12. Following the Week 12 visit, participants who completed Part 1 of the study received open-label 8 mg/kg tocilizumab through Week 208.
  Interventions: Drug: Placebo
- Part 1: Tocilizumab (Experimental): Participants received intravenous infusions of 8 mg/kg tocilizumab once every 4 weeks until Week 12. Following the Week 12 visit, participants who completed Part 1 of the study received open-label 8 mg/kg tocilizumab through Week 208.
  Interventions: Biological: tocilizumab
- Part 2: Placebo (Placebo Comparator): Participants received intravenous infusions of placebo once every 4 weeks until Week 24. Participants who did not attain an ASsessment in Ankylosing Spondylitis-20 (ASAS20) response at Week 16 were, at the investigator's discretion, eligible to receive open-label escape therapy consisting of 8 mg/kg tocilizumab. After Week 24, participants were to receive open-label treatment with 8 mg/kg tocilizumab every 4 weeks until Week 104. At the completion of Week 104, all Part 2 participants were to receive tocilizumab 8 mg/kg in the common open-label extension phase, however the study was terminated prior to any participants reaching this stage.
  Interventions: Drug: Placebo
- Part 2: Tocilizumab 4 mg/kg (Experimental): Participants received intravenous infusions of 4 mg/kg tocilizumab once every 4 weeks until Week 24. Participants who did not attain an ASAS20 response at Week 16 were, at the investigator's discretion, eligible to receive open-label escape therapy consisting of 8 mg/kg tocilizumab. After Week 24, participants were to receive open-label treatment with 8 mg/kg tocilizumab every 4 weeks until Week 104. At the completion of Week 104, all Part 2 participants were to receive tocilizumab 8 mg/kg in the common open-label extension phase, however the study was terminated prior to any participants reaching this stage.
  Interventions: Biological: tocilizumab
- Part 2: Tocilizumab 8 mg/kg (Experimental): Participants received intravenous infusions of 8 mg/kg tocilizumab once every 4 weeks until Week 24. Participants who did not attain an ASAS20 response at Week 16 were, at the investigator's discretion, eligible to receive open-label escape therapy consisting of 8 mg/kg tocilizumab. After Week 24, participants were to receive open-label treatment with 8 mg/kg tocilizumab every 4 weeks until Week 104. At the completion of Week 104, all Part 2 participants were to receive tocilizumab 8 mg/kg in the common open-label extension phase, however the study was terminated prior to any participants reaching this stage.
  Interventions: Biological: tocilizumab

INTERVENTIONS:
Biological: tocilizumab — Administered intravenously (iv) every 4 weeks
  Other Names: RoActemra/Actemra
  Arms: Part 1: Tocilizumab; Part 2: Tocilizumab 4 mg/kg; Part 2: Tocilizumab 8 mg/kg
Drug: Placebo — Placebo to tocilizumab administered intravenously every 4 weeks
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the safety and efficacy of RoActemra/Actemra (tocilizumab) in patients with ankylosing spondylitis (AS) who have failed treatment with non-steroidal anti-inflammatory drugs and are naïve to tumor necrsos factor (TNF) antagonist therapy. In Part 1 of the study, patients will be randomized to receive either RoActemra/Actemra 8 mg/kg intravenously (IV) or placebo every 4 weeks for 12 weeks. In Part 2, patients will be randomized to receive RoActemra at either 8 mg/kg or 4 mg/kg IV or placebo every 4 weeks for 24 weeks. The double-blind treatment period will be followed by open-label treatment with RoActemra/Actemra 8 mg/kg iv every 4 weeks until Week 208 for all patients. Anticipated time on study treatment is 208 weeks.

DETAILED DESCRIPTION:
This study was planned as a Phase II/III seamless, multicenter, randomized, double-blind, placebo-controlled study in patients with AS who were naïve to TNF antagonist therapy. The study consisted of 2 parts, each preceded by a screening visit and followed by a common open-label extension phase. Recruitment into Part 2 commenced after completion of enrollment for Part 1.

Part 1 was designed as a Phase II study exploring the efficacy and safety of tocilizumab therapy versus placebo. Part 1 was intended to determine whether Part 2 of the study would continue, based on a Week 12 analysis.

Part 2 was designed to provide pivotal Phase III efficacy and safety data for tocilizumab in patients with AS. Approximately 400 patients were to be enrolled. Once randomization into Part 1 was complete, randomization into Part 2 of the study was to be initiated.

Based on the results of the Week 12 Part 1 analyses of the primary endpoint (ASAS20) and secondary endpoints, and in consideration of all available safety data, a benefit/risk assessment was made and it was decided to halt the study because of lack of overall efficacy. Most patients did not complete the 24-week double-blind treatment period in Part 2.

ELIGIBILITY:
Inclusion Criteria

* Adult patients, ≥ 18 years of age
* Ankylosing Spondylitis as defined by the modified New York criteria for ≥ 3 months prior to baseline
* Active disease at screening and baseline (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] ≥4.0, spinal pain visual analog scale [VAS] ≥40)
* Inadequate response or intolerant to 1 or more previous non-steroidal anti-inflammatory drugs (NSAIDs)
* Traditional disease-modifying anti-rheumatic drugs (DMARDs) must be withdrawn for at least 4 weeks prior to baseline (methotrexate, sulfasalazine and hydroxychloroquine or chloroquine may be allowed if at stable dose for at least 4 weeks prior to baseline)
* Oral corticosteroids (≥ 10 mg/day prednisone or equivalent) and NSAIDs/COX-2 inhibitors must be at stable dose for at least 4 weeks prior to baseline

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months after randomization
* Total ankylosis of spine (as determined by investigator)
* Inflammatory rheumatic disease other than ankylosing spondylitis
* Active, acute uveitis at baseline
* Treatment with tumor necrosis factor (TNF) antagonist therapy at any time prior to baseline
* Intra-articular or tendon injections or parenteral corticosteroids within 4 weeks prior to screening
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infection
* History of or currently active primary or secondary immunodeficiency
* Body weight > 150 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (114):
- United States (15):
  - Huntington Beach, California
  - Aventura, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Idaho Falls, Idaho
  - Wichita, Kansas
  - Cumberland, Maryland
  - Saint Claire Shores, Michigan
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Duncansville, Pennsylvania
  - Hickory Grove, South Carolina
  - Houston, Texas
- Australia (7):
  - Adelaide
  - Heidelberg
  - Hobart
  - Malvern East
  - Maroochydore
  - Sydney
  - Woodville
- Belgium (4):
  - Brussels
  - Kortrijk
  - Liège
  - Yvoir
- Brazil (3):
  - Cuiabá
  - Goiânia
  - São Paulo
- Bulgaria (4):
  - Plovdiv
  - Rousse
  - Sevlievo
  - Sofia
- Canada (11):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Kitchener, Ontario
  - Mississauga, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec
  - Trois-Rivières, Quebec
- Czechia (8):
  - Bruntál
  - Hlučín
  - Olomouc
  - Prague
  - Praha 4 Nusle
  - Sokolov
  - Uherské Hradiště
  - Zlín
- France (8):
  - Besançon
  - Boulogne-Billancourt
  - Créteil
  - Grenoble
  - Montpellier
  - Paris
  - Strasbourg
  - Toulouse
- Germany (5):
  - Berlin
  - Cologne
  - Gommern
  - Hanover
  - Würzburg
- India (6):
  - Ahmedabad
  - Bangalore
  - Hyderabad
  - Jaipur
  - New Delhi
  - Secunderabad
- Italy (7):
  - Ferrara
  - Florence
  - Monserrato
  - Prato
  - Reggio Emilia
  - Roma
  - Siena
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (7):
  - Bydgoszcz
  - Krakow
  - Lublin
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- Russia (4):
  - Kazan'
  - Moscow
  - Voronezh
  - Yaroslavl
- Slovakia (2):
  - Košice
  - Piešťany
- South Africa (4):
  - Cape Town
  - Durban
  - Pretoria
  - Stellenbosch
- Spain (7):
  - A Coruña
  - Barcelona
  - Córdoba
  - Lugo
  - Madrid
  - Oviedo
  - Sabadell
- United Kingdom (9):
  - Basingstoke
  - Bath
  - Cannock
  - Greenock
  - Leeds
  - London
  - Salford
  - Stoke-on-Trent
  - Wigan

REFERENCES:
- [Derived] Sieper J, Porter-Brown B, Thompson L, Harari O, Dougados M. Assessment of short-term symptomatic efficacy of tocilizumab in ankylosing spondylitis: results of randomised, placebo-controlled trials. Ann Rheum Dis. 2014 Jan;73(1):95-100. doi: 10.1136/annrheumdis-2013-203559. Epub 2013 Jun 13. PMID 23765873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part 1, patients were randomized in a 1:1 ratio to placebo or tocilizumab (TCZ) 8 mg/kg. In Part 2, patients were randomized in a 2:1:1 ratio to TCZ 8 mg/kg, TCZ 4 mg/kg, or placebo, respectively. Due to the early stopping of the study and limitations in available data the TCZ dose groups in Part 2 were combined.
Groups:
- Part 1: Placebo: Participants received intravenous infusions of placebo once every 4 weeks until Week 12. Following the Week 12 visit, participants were to receive open-label 8 mg/kg tocilizumab through Week 208 in the common open-label extension phase.
- Part 1: Tocilizumab: Participants received intravenous infusions of 8 mg/kg tocilizumab once every 4 weeks until Week 12. Following the Week 12 visit, participants were to receive open-label 8 mg/kg tocilizumab through Week 208 in the common open-label extension phase.
- Part 2: Placebo: Participants received intravenous infusions of placebo once every 4 weeks until Week 24. Participants who did not attain an ASsessment in Ankylosing Spondylitis-20 (ASAS20) response at Week 16 were eligible to receive open-label escape therapy consisting of 8 mg/kg tocilizumab. After Week 24, participants were to receive open-label treatment with 8 mg/kg tocilizumab every 4 weeks until Week 104. At the completion of Week 104, all Part 2 participants were to receive tocilizumab 8 mg/kg in the common open-label extension phase.
- Part 2: Tocilizumab: Participants received intravenous infusions of 4 mg/kg or 8 mg/kg tocilizumab once every 4 weeks until Week 24. Participants who did not attain an ASAS20 response at Week 16 were eligible to receive open-label escape therapy consisting of 8 mg/kg tocilizumab. After Week 24, participants were to receive open-label treatment with 8 mg/kg tocilizumab every 4 weeks until Week 104. At the completion of Week 104, all Part 2 participants were to receive tocilizumab 8 mg/kg in the common open-label extension phase.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Started | 51 | 51 | 51 | 153
Treated | 51 | 51 | 51 | 152
Escape or Switched to Tocilizumab | 51 | 0 | 6 | 0
Completed 12 Weeks Treatment | 50 | 48 | 12 | 59
Completed 24 Weeks Treatment | 19 | 28 | 3 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 51 | 51 | 51 | 153

BASELINE CHARACTERISTICS:
Groups:
- Combined Placebo: Participants in Part 1 and Part 2 who received intravenous infusions of placebo once every 4 weeks.
- Combined Tocilizumab: Participants randomized in Part 1 and Part 2 to receive intravenous infusions of 4 mg/kg (in Part 2 only) or 8 mg/kg tocilizumab once every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Combined Placebo | Combined Tocilizumab | Total
Number analyzed (Participants) | 102 | 203 | 305
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for all participants who received at least one tocilizumab/placebo infusion.
  years | 41.2 (11.33) | 40.4 (11.42) | 40.7 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 53 | 82
  Male | 73 | 150 | 223
Age - Part 1 population [Mean (Standard Deviation); unit: years] — Demographic data for the Part 1 population: Placebo = 51 participants, Tocilizumab = 51 participants, total = 102 participants.
  years | 42.7 (12.64) | 41.6 (11.22) | 42.1 (11.91)
Gender - Part 1 Population [Number; unit: participants] — Demographic data for the Part 1 population: Placebo = 51 participants, Tocilizumab = 51 participants, total = 102 participants.
  participants
    Female | 11 | 15 | 26
    Male | 40 | 36 | 76

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Achieving a 20% Improvement in Assessment in Ankylosing Spondylitis (ASAS20) at Week 12
Description: ASAS is composed of four domains. To achieve an ASAS20 response required improvement of ≥20% and ≥ 1 unit (10 mm) in at least 3 domains and no worsening of ≥ 20 % and ≥ 1 unit (10 mm) in the remaining domain.
  * The patient's global assessment of current disease status, measured on a 100 mm visual analog scale (VAS), from symptom-free / no AS symptoms (0) to maximum AS disease severity (100).
  * The patient's overall assessment of the severity of spinal pain based on responses to 2 questions assessed on a 100 mm VAS, from no pain (0) to most severe pain (100). The spinal pain score is the mean of these 2 questions.
  * The function component was measured by the Bath Ankylosing Spondylitis Functional Index (BASFI). The patient provides self-assessment of 10 questions on a 100 mm VAS. The BASFI score is the mean of these values.
  * The inflammation component of the ASAS was determined by the mean of questions 5 and 6 of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI).
Time Frame: Baseline and Week 12
Population: Intent-to-treat (ITT) population included all patients who were randomized into the study and received at least one tocilizumab/placebo infusion.
  If the response at the 12-week visit could not be determined due to early withdrawal or missing data then the patient was considered a non-responder.
Measure: Number; unit: percentage of participants
Groups:
- Part 1: Placebo: Participants received intravenous infusions of placebo once every 4 weeks until Week 12.
- Part 1: Tocilizumab: Participants received intravenous infusions of 8 mg/kg tocilizumab once every 4 weeks until Week 12.
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab
Number analyzed (Participants) | 51 | 51
percentage of participants | 27.5 | 37.3

2. Secondary Outcome: Part 2: Percentage of Participants Achieving a 20% Improvement in Assessment in Ankylosing Spondylitis (ASAS20) at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Intent-to-treat (ITT) population. The analysis only includes assessments while the patient was receiving double blind medication, and occurred prior to both withdrawal and the 15 July 2011 (date at which all patients were unblinded). Patients who withdrew or escaped are considered as non-responders until week 24.
Measure: Number; unit: percentage of participants
Groups:
- Part 2: Placebo: Participants received intravenous infusions of placebo once every 4 weeks.
- Part 2: Tocilizumab: Participants received intravenous infusions of 4 mg/kg or 8 mg/kg tocilizumab once every 4 weeks.
Arm/Group | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 49 | 101
percentage of participants | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants Who Achieved a Value <2 in Each of the 4 ASAS Parameters at Week 12
Description: Assessment in Ankylosing Spondylitis (ASAS) is composed of four domains.
  * The patient's global assessment of current disease status, measured on a 100 mm visual analog scale (VAS), from symptom-free / no AS symptoms (0) to maximum AS disease severity (100).
  * The patient's overall assessment of the severity of spinal pain based on responses to 2 questions assessed on a 100 mm VAS, from no pain (0) to most severe pain (100). The spinal pain score is the mean of these 2 questions.
  * The function component was measured by the Bath Ankylosing Spondylitis Functional Index (BASFI), the mean of 10 self-assessment questions on a 100 mm VAS.
  * The inflammation component of the ASAS was determined by the mean of questions 5 and 6 of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI).
  Each of the above 4 domains are measured on a scale from 0-100 mm, but reported on a 0-10 cm scale. A score of less than 2 units (20 mm) in each domain is defined as partial remission.
Time Frame: Week 12
Population: Intent-to-treat. If the response at the Week 12 visit could not be determined due to early withdrawal or missing data then the patient is considered a non-responder. The analysis was not performed for participants in Part 2 due to premature study termination.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 51 | 0 | 0
percentage of participants | 2.0 | 0.0 |  |

4. Secondary Outcome: Percentage of Participants Achieving a 40% Improvement in Assessment in Ankylosing Spondylitis (ASAS40) at Week 12
Description: ASAS is composed of four domains. To achieve an ASAS40 response required improvement of ≥40% and ≥ 2 units (20 mm) in at least 3 domains and no worsening at all in the remaining domain.
  * The patient's global assessment of current disease status, measured on a 100 mm visual analog scale (VAS), from symptom-free / no AS symptoms (0) to maximum AS disease severity (100).
  * The patient's overall assessment of the severity of spinal pain based on responses to 2 questions assessed on a 100 mm VAS, from no pain (0) to most severe pain (100). The spinal pain score is the mean of these 2 questions.
  * The function component was measured by the Bath Ankylosing Spondylitis Functional Index (BASFI). The patient provides self-assessment of 10 questions on a 100 mm VAS. The BASFI score is the mean of these values.
  * The inflammation component of the ASAS was determined by the mean of questions 5 and 6 of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI).
Time Frame: Baseline and Week 12
Population: Intent-to-treat (ITT) population. If the response at the Week 12 visit could not be determined due to early withdrawal or missing data then the patient is considered a non-responder. The analysis was not performed for participants in Part 2 due to premature study termination.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 51 | 0 | 0
percentage of participants | 19.6 | 11.8 |  |

5. Secondary Outcome: Part 2: Percentage of Participants Achieving a 40% Improvement in Assessment in Ankylosing Spondylitis (ASAS40) at Week 24
Description: as for outcome 4
Time Frame: Baseline and Week 24
Population: Intent-to-treat (ITT), Part 2 study population. This analysis was not performed due to premature study termination.
Arm/Group | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI is a patient-administered assessment of 6 parameters specific to AS. The following parameters were assessed on a 100-mm horizontal visual analogue: fatigue, spinal pain, peripheral arthritis, enthesitis, intensity of morning stiffness, and duration of morning stiffness. For questions 1 to 5, the left-hand extreme of the line (0) represents "none" (symptom-free) and the right-hand extreme (100) represents "very severe" (maximum severity). For question 6, a time axis was used, with the left-hand extreme of the line representing "0 hours" and the right-hand extreme representing "2 or more hours". The BASDAI score was calculated as follows:
  BASDAI = [Q1 + Q2 + Q3 + Q4 + (Q5 + Q6)/2]/5. The total score is tabulated on a scale from 0 (best) to 10 cm (worst).
Time Frame: Baseline and Week 12
Population: Intent-to-treat population where data were available.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 51 | 51 | 152
cm
  Baseline [N=51, 51, 51, 152] | 6.77 (1.322) | 6.62 (1.327) | 6.86 (1.506) | 6.41 (1.527)
  Week 12 [N=51, 48, 20, 53] | 5.65 (2.042) | 5.64 (1.833) | 6.20 (1.900) | 5.39 (2.183)
  Change from Baseline [N=51, 48, 20, 53] | -1.12 (1.991) | -1.02 (1.813) | -0.53 (1.637) | -1.17 (1.919)

7. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) is an assessment of function in AS patients. The participant provides their assessment of their ability to perform 10 activities on a 100 mm horizontal visual analog scale (VAS) ranging from 0 (easy) to 100 (impossible). The BASFI score is the mean of these values and is tabulated on a 0 (best) to 10 (worst) cm scale.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population for whom data were available. The analysis was not performed for participants in Part 2.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 51 | 0 | 0
cm
  Baseline [N=51,51] | 5.60 (2.071) | 6.24 (2.069) |  |
  Week 12 [N=51, 48] | 4.84 (2.257) | 5.55 (2.004) |  |
  Change from Baseline [N=51, 48] | -0.76 (1.660) | -0.73 (1.736) |  |

8. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: The Bath Ankylosing Spondylitis Metrology Index linear function is a combined index of 5 clinical measurements (performed by the Joint Assessor) which reflect axial mobility in the AS patient. The measurements to assess mobility are:
  1. Tragus-to-wall;
  2. Modified Schober (lumbar flexion);
  3. Cervical rotation;
  4. Lateral spinal flexion;
  5. Intermalleolar distance.
  The BASMI linear result is the average of the 5 assessments and ranges from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their AS.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population where data were available. The analysis was not performed for participants in Part 2 due to premature study termination.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 51 | 0 | 0
scores on a scale
  Baseline [N=50, 47] | 4.35 (1.604) | 4.58 (1.772) |  |
  Week 12 [N=50, 47] | 4.29 (1.682) | 4.40 (1.943) |  |
  Change from Baseline [N=50, 46] | -0.06 (0.832) | -0.21 (1.197) |  |

9. Secondary Outcome: Change From Baseline in C-Reactive Protein
Description: Levels of C-reactive protein (CRP) were measured from blood samples taken at Baseline and at Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 51 | 0 | 0
mg/dL
  Baseline [N=51, 51] | 1.75 (1.850) | 1.62 (2.248) |  |
  Week 12 [N=50, 48] | 1.58 (1.733) | 0.36 (1.008) |  |
  Change from Baseline [N=50, 48] | -0.17 (1.005) | -1.34 (2.442) |  |

10. Secondary Outcome: Part 2: Area Under the Plasma Concentration Versus Time Curve of Tocilizumab
Description: Area under the plasma concentration versus time curve (AUC) of tocilizumab at steady state after 12 weeks of treatment.
Time Frame: Week 12, pre-dose and at the end of infusion, on the 2nd and 7th day of Week 12, 14 days post-dose (Week 14) and 28 days post-dose (pre-dose of Week 16 infusion).
Population: Due to premature study termination pharmacokinetic parameters were not analyzed.
Arm/Group | Part 2: Tocilizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Part 2: Peak Plasma Concentration of Tocilizumab
Description: The peak plasma concentration (Cmax) of tocilizumab at steady state after 12 weeks of treatment.
Time Frame: as for outcome 10
Population: Due to premature study termination pharmacokinetic parameters were not analyzed.
Arm/Group | Part 2: Tocilizumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Part 2: Elimination Half-life of Tocilizumab
Description: Elimination half-life of tocilizumab at steady state after 12 weeks of treatment.
Time Frame: as for outcome 10
Population: Due to premature study termination pharmacokinetic parameters were not analyzed.
Arm/Group | Part 2: Tocilizumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Part 2: Clearance of Tocilizumab
Description: Clearance of tocilizumab at steady state after 12 weeks of treatment.
Time Frame: as for outcome 10
Population: Due to premature study termination pharmacokinetic parameters were not analyzed.
Arm/Group | Part 2: Tocilizumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Part 2: Volume of Distribution of Tocilizumab
Description: Volume of distribution of tocilizumab at steady state after 12 weeks of treatment.
Time Frame: as for outcome 10
Population: Due to premature study termination pharmacokinetic parameters were not analyzed.
Arm/Group | Part 2: Tocilizumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Change From Baseline in the Level of Interleukin-6
Description: Interleukin-6 levels were measured from blood samples taken pre-dose at Baseline and after 12 weeks of treatment.
  The analysis was not performed for participants in Part 2 due to premature study termination.
Time Frame: Baseline and Week 12
Population: Pharmacokinetic (PK) Population: All patients who received at least one tocilizumab infusion and had at least one PK and pharmacodynamic sample. Only patients with available data at each time point are included (indicated by N). Patients who did not receive their Week 8 dose were excluded.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part 1: Tocilizumab | Part 2: Tocilizumab
Number analyzed (Participants) | 44 | 0
pg/mL
  Baseline [N=41] | 10 (11.8) |
  Week 12 [N=40] | 78 (61.5) |
  Change from Baseline [N=37] | 67 (58.3) |

16. Secondary Outcome: Change From Baseline in Level of Soluble Interleukin-6 Receptor
Description: Soluble Interleukin-6 receptor levels were measured from blood samples taken pre-dose at Baseline and after 12 weeks of treatment.
  The analysis was not performed for participants in Part 2 due to premature study termination.
Time Frame: Baseline and Week 12
Population: Pharmacokinetic Population: All patients who received at least one tocilizumab infusion and had at least one pharmacokinetic and pharmacodynamic sample. Only those patients with available data at each time point are included in the analysis (indicated by N). Patients who did not receive their week 8 dose were excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Tocilizumab | Part 2: Tocilizumab
Number analyzed (Participants) | 44 | 0
ng/mL
  Baseline [N=41] | 42 (11.5) |
  Week 12 [N=40] | 536 (173.1) |
  Change from Baseline [N=37] | 496 (173.9) |

17. Secondary Outcome: Number of Participants With Anti-tocilizumab Antibodies
Description: A positive anti-tocilizumab antibody result was defined as a negative assay result at Baseline and a positive post-baseline screening assay with positive confirmation or neutralizing assay at the same visit.
Time Frame: From Baseline until end of study (a maximum treatment duration of 40 weeks).
Population: All patients treated with tocilizumab and screened for anti-tocilizumab antibodies at any timepoint.
Measure: Number; unit: participants
Groups:
- All Tocilizumab: Participants who received intravenous infusions of 4 mg/kg or 8 mg/kg tocilizumab once every 4 weeks in either Part 1 or Part 2, including participants randomized to placebo who switched or escaped to tocilizumab treatment.
Arm/Group | All Tocilizumab
Number analyzed (Participants) | 257
participants | 4

18. Primary Outcome: Part 2: Percentage of Participants Achieving a 20% Improvement in Assessment in Ankylosing Spondylitis (ASAS20) at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 51 | 119
percentage of participants | 7.8 | 9.2

19. Secondary Outcome: Part 2: Radiographic Change According to the Modified Stoke Ankylosing Spondylitis Spinal Score (mSASSS)
Description: Radiographs were to be assessed using the modified Stoke Ankylosing Spondylitis Spinal Score (mSASSS). The mSASSS is a four-point scoring system for lateral radiographs of the lumbar and cervical spine and has been shown to reliably track disease progression over time, where:
  * 0 = No abnormality;
  * 1 = Erosion, sclerosis, or squaring;
  * 2 = Syndesmophyte;
  * 3 = Total bony bridging at each site.
Time Frame: Baseline and Week 104
Population: This outcome measure was not analyzed due to premature study termination.
Arm/Group | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Part 2: Percentage of Participants With a Reduction of Magnetic Resonance Imaging (MRI) Proven Spinal Inflammation
Description: Magentic resonance imaging of the axial skeleton was to be performed at Baseline and Week 24. MRI scans will be evaluated using the ankylosing spondylitis spinal MRI activity (ASspiMRI-a) score, grading activity (0-6) per vertebral unit in 23 units.
Time Frame: Baseline and Week 24
Population: Due to premature study termination this outcome measure was not analyzed.
Arm/Group | Part 2: Placebo | Part 2: Tocilizumab
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Part 1: The Number of Participants With Adverse Events
Description: A serious adverse event (AE) is any event that is fatal, life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant or requires intervention to prevent one or other of the outcomes listed above. The intensity of each AE was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.02. A severe AE was any event of Grade 4 (life-threatening consequences; urgent intervention indicated) or 5 (death related to AE).
Time Frame: Up to 40 weeks
Population: The safety analysis population included all patients who received at least one tocilizumab/placebo infusion and had at least one postdose safety assessment. Patients were assigned to treatment groups as treated for analysis.
Measure: Number; unit: participants
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab
Number analyzed (Participants) | 51 | 51
participants
  Any adverse event | 27 | 30
  Serious adverse event | 0 | 2
  Death | 0 | 0
  Withdrawals due to AE | 0 | 0
  Severe AE | 0 | 0

ADVERSE EVENTS:
Groups:
- Part 2: Placebo: Participants received intravenous infusions of placebo once every 4 weeks. AEs reported only until participants escaped or switched to tocilizumab.
- All Tocilizumab: Participants who received intravenous infusions of 4 mg/kg or 8 mg/kg tocilizumab once every 4 weeks in either Part 1 or Part 2. This group includes participants randomized to placebo who switched or escaped to tocilizumab treatment for whom adverse events are reported after the start of treatment with tocilizumab.
Arm/Group | Part 1: Placebo | Part 1: Tocilizumab | Part 2: Placebo | All Tocilizumab
Serious Adverse Events (participants affected / at risk) | 0/51 | 2/51 | 0/51 | 11/260
Other Adverse Events (participants affected / at risk) | 1/51 | 3/51 | 1/51 | 8/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=51) | Part 1: Tocilizumab (N=51) | Part 2: Placebo (N=51) | All Tocilizumab (N=260)
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Bursitis infective staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=51) | Part 1: Tocilizumab (N=51) | Part 2: Placebo (N=51) | All Tocilizumab (N=260)
Hypertension (Vascular disorders) | 1 | 3 | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.